CLINICAL TRIAL: NCT00481000
Title: Dialectical Cognitive Traumatherapy (DCT) on Patients With Severe Posttraumatic Stress Disorder Following Sexual Abuse - A Randomised Controlled Trial
Brief Title: Dialectical Cognitive Traumatherapy (DCT) on Patients With Severe PTSD Following Sexual Abuse
Acronym: PASA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Prof. Dr. Martin Bohus, Central Institute of Mental Health, Psychosomatic Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PASA-0230
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Dialectical Cognitive Therapy; Clinical Psychology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): Waitlist; Treatment as usual
  Interventions: Behavioral: Dialectical Cognitive Therapy

INTERVENTIONS:
Behavioral: Dialectical Cognitive Therapy — Dialectical Behavior Therapy in Combination with Traumafocused CBT

SUMMARY:
The purpose of this study is to determine whether Dialectical Cognitive Traumatherapy is effective in the treatment of severe and chronic Posttraumatic Stress Disorder (PTSD) following childhood sexual abuse.

DETAILED DESCRIPTION:
Most studies on psychological treatments for PTSD exclude patients with severe, co-occurring psychopathology. We designed a new treatment (Dialectical Cognitive Trauma Therapy, or DCT) specifically to treat these patients. DCT includes elements of emotion regulation, mindfulness exercises, cognitive and exposure treatment, as well as new elements. This randomized controlled study evaluates the effect of inpatient DCT on these patients.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Minimum age of 17
* Childhood sexual abuse
* Posttraumatic Stress Disorder (criteria of SCID)
* At least one of the following diagnoses: Anorexia Nervosa, or Bulimia Nervosa, or substance abuse, or substance dependence, or major depression or at least 4 out of 9 criteria for Borderline Personality Disorder

Exclusion Criteria:

* Diagnosis of schizophrenia
* Mental retardation
* Body Mass Index lower than 16.5
* Acute delirium
* Perilous selfharming behaviour during the last 4 month
* Suicide attempt with the distinct intention to die during the last 4 month
* Unstability (e.g. homelessness, acute victimisation by offender)
* Pretreatment by DCT

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-12 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptoms (CAPS, SCID, PDS, IESR) | 1.5 years

SECONDARY OUTCOMES:
general psychopathology | 1.5 years
change of pain threshold | 1.5 years
fMRI: activity of the amygdala | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Regina Steil, PhD, Study Director — Central Institute of Mental Health; Martin Bohus, PhD, Study Chair — Central Institute of Mental Health; Anne S Dyer, PhD, Principal Investigator — Central Institute of Mental Health
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Gorg N, Priebe K, Bohnke JR, Steil R, Dyer AS, Kleindienst N. Trauma-related emotions and radical acceptance in dialectical behavior therapy for posttraumatic stress disorder after childhood sexual abuse. Borderline Personal Disord Emot Dysregul. 2017 Jul 13;4:15. doi: 10.1186/s40479-017-0065-5. eCollection 2017. PMID 28717512